CLINICAL TRIAL: NCT04721587
Title: Effectiveness of Virtual Reality as a Pain and Anxiety Distraction Strategy on Office Hysteroscopy
Brief Title: Virtual Reality for Pain and Anxiety Distraction Strategy on Office Hysteroscopy
Acronym: VRPAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Psious (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-VIR-2019-75
Record Dates: First submitted 2020-12-11; First posted 2021-01-22 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2021-01

CONDITIONS: Pain, Acute; Anxiety
Keywords: Hysteroscopy; Pain; Virtual Reality; Anxiety
MeSH Terms: conditions — Acute Pain; Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Office hysteroscopy performed as the standard of care of our Hospital
- Virtual Reality (Experimental): Office hysteroscopy with the use of VR environment (preprocedure and during procedure)
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — The patients of the VR Group will be subjected to the same hysteroscopy technique as the Standard of Care Group, but additionally a VR device will be applied where a distraction VR environment ("Underwater Game") will be reproduced during the exploration
  Arms: Virtual Reality

SUMMARY:
Hysteroscopy is a minimally invasive endoscopic technique that allows direct visualization of the uterine cavity and constitutes the gold standard for the diagnosis and treatment of most intrauterine pathology, such as heavy menstrual bleeding, fibroids, endometrial polyps, uterine malformations, etc. The "see and treat" strategy allows diagnosis and treatment in the same surgical act, and gives the technique a high resolution capacity, reducing the number of procedures the patient must undergo. The technological development of instruments has made it possible to have small-caliber endoscopic systems that have made this technique possible in an outpatient setting. Outpatient management allows patients to avoid the possible risks and inconveniences associated with the surgical environment, such as the waiting list and the need for anesthesia, as well as an earlier return to their activities of daily life. Despite the high resolution rates, a not inconsiderable percentage of women experience anxiety or pain during outpatient hysteroscopy, and this is the leading cause of treatment failure. In order to improve the tolerance and comfort of the patient, the usefulness of various strategies, both pharmacological and non-pharmacological, has been evaluated for pain reduction, with different results.

Virtual Reality (VR) has been used successfully to reduce perceived pain in various procedures such as chronic pain, burns, dental processes, chronic pruritus or venipuncture. There is no published study to our knowledge that evaluates the usefulness of VR in reducing the levels of anxiety and pain perceived during a hysteroscopic procedure.

The working hypothesis to be evaluated with this study is that the use of a VR device with reproduction of relaxing and distraction environments reduces the perception of pain and anxiety of the patient during an outpatient hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years
* Understand and accept the study procedures
* Sign the informed consent.
* Indication of outpatient hysteroscopy according to the care protocols of the center
* Not taking drugs for the treatment of anxiety.

Exclusion Criteria:

* Not being able to understand the nature of the study and / or the procedures to be followed
* Not signing the informed consent
* Be under the age of 18
* Pregnancy
* Being diagnosed with anxiety disorder or being treated with anxiolytics
* Patients suffering from vertigo
* Patients with epilepsy
* Active ear infection
* Patients with diagnosed hypertension
* Patients with cardiovascular disease
* Patients with psychosis or severe mental illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Pain score | Intraprocedure
  Decrease of 1 point or more in the level of pain measured by an 11-point visual analog scale, a validity scale that comprises 11 consecutive values from 0 to 10, with "0" corresponding to no pain and "10" to worst pain imaginable.

SECONDARY OUTCOMES:
Heart Rate | Intraprocedure
  Changes in basal Heart Rate, maximum Heart Rate, mean Heart Rate, and final Heart Rate.
Blood Pressure | Intraprocedure
  Changes in pre and postprocedure blood pressure
Skin conductace | Intraprocedure
  Change between basal and maximum skin conductance levels during pocedure measured by a small sensor placed on two hand fingers. Skin conductance depends directly on the state of relaxation or stress, making it a commonly used and very precise stress indicator.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Estadella Tarriel, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain